CLINICAL TRIAL: NCT03680898
Title: Prospective Study for Clinical Validation of the Molecular-Based GenePOC Carba Assay for the Detection and Differentiation of Carbapenemase Genes of Gram-negative Bacteria (blaIMP, blaKPC, blaNDM, blaOXA-48-like and blaVIM) in Rectal Swab Samples From Patients Suspected of Being Colonized. The Targeted Organisms Are Enterobacteriaceae, Acinetobacter Baumannii, and Pseudomonas Aeruginosa.
Brief Title: Clinical Validation of the Molecular-Based GenePOC Carba Assay for the Detection and Differentiation of Carbapenemase Genes in Rectal Swab Samples.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Meridian Bioscience, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: GPC04-003
Record Dates: First submitted 2018-09-20; First posted 2018-09-21 (Actual); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Carbapenem-Resistant Enterobacteriaceae
Keywords: Carbapenem; rectal swab; infectious disease; infection
MeSH Terms: conditions — Communicable Diseases; Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- revogene Testing (Experimental): The swab will be used for the testing on the revogene using the GenePOC Carba assay.
  Interventions: Device: Rectal swab collection
- Reference Method (Active Comparator): The other swab will be used in the Reference Method.
  Interventions: Device: Rectal swab collection

INTERVENTIONS:
Device: Rectal swab collection — Patient will provide a rectal swab by following hospital-provided instructions.

SUMMARY:
The primary purpose of this clinical investigation is to establish the performance of the GenePOC Carba assay on the revogene. This will be achieved by comparing the test to a conventional method for detection of Carbapenemase Producing Organisms (CPOs) in rectal swab samples.

DETAILED DESCRIPTION:
The GenePOC Carba assay will be performed using the revogene instrument. The revogene instrument, used in conjunction with appropriate reagents, is capable of automated cell lysis, dilution of nucleic acids from multiple sample types as well as automated amplification and detection of target nucleic acid sequences.

The GenePOC Carba assay reagents kits consist of:

1. Sample Buffer Tube (SBT)
2. Disposable Transfer Tool (DTT)
3. Disposable microfluidic cartridges (PIE)

The test is performed using the revogene™. The revogene automates sample homogenization, sample dilution, cells lysis, DNA amplification, and detection of the amplified PCR products. User intervention is only required for discharging the patient sample into the Sample Buffer Tube (SBT), transferring the sample into the PIE, and loading/unloading the PIEs into the revogene carousel.

A dual swab sample is collected when ICF is signed by patient. One of the swab is transferred into the SBT and vortexed. Sample is then transferred to the GenePOC Carba PIE. The PIE is then automatically processed by the revogene. On completion of a run, the user removes the processed PIEs from the instrument and discards them according to local biological waste management procedures.

One revogene will be allocated per site. The purpose of this clinical trial is to enroll sufficient patients from up to 14 Clinical Centers to meet regulatory requirements, based on the Reference Method final results.

ELIGIBILITY:
Inclusion Criteria:

* Samples from patients who were previously diagnosed to be infected with CPOs, or were identified per hospital policies as being suspected or are at risk for CPO infection;
* Patient that signed the approved Informed Consent Form (if applicable)
* Patient older than 2 years of age (>24.0 months)
* Only one (1) compliant sample per patient is allowed

Exclusion Criteria:

* Patient/sample not meeting inclusion criteria above

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2019-02-12 (Actual); Primary Completion 2023-05-31 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Performance characteristics : Clinical sensitivity (true positive rate) in comparison to the Reference Method | up to 3 months
  To establish the performance characteristics of the GenePOC Carba assay for its use in determining the presence of CPO/CPE in rectal swab samples obtained from patients suspected of being infected, or considered at risk.
  Sensitivity will be estimated as the proportion of positives that are correctly identified by the Carba assay when compared to the Reference Method.
Performance characteristics : clinical specificity (true negative rate) in comparison to the Reference Method | up to 3 months
  To establish the performance characteristics of the GenePOC Carba assay for its use in determining the presence of CPO/CPE in rectal swab samples obtained from patients suspected of being infected, or considered at risk.
  Sensitivity will be estimated as the proportion of positives that are correctly identified by the Carba assay when compared to the Reference Method.

CONTACTS AND LOCATIONS:
Overall Officials: Keith Chiasson, PhD, Study Director — Meridian Bioscience, Inc.
Locations (3):
- United States (2):
  - Indiana University and Purdue University Institutions, Indianapolis, Indiana
  - Henry Ford Health System, Detroit, Michigan
- Mount Sinai Hospital Joseph and Wolf Lebovic Health Complex, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No